CLINICAL TRIAL: NCT07133620
Title: The Effect of Transcutaneous Electrical Acupoint Stimulation on Postoperative Gastrointestinal Dysfunction After Urological Laparoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Yang Bin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FirstAHXiamenU-YB-4
Record Dates: First submitted 2025-08-09; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Gastrointestinal Dysfunction (POGD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Sham Comparator)
  Interventions: Device: Sham transcutaneous Electrical Acupoint Stimulation
- TEAS group (Experimental)
  Interventions: Device: Transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — Before the operation, the patient received transcutaneous electrical acupoint stimulation (TEAS) at bilateral Zusanli (ST 36), Neiguan (PC 6), and Ciliao (BL 32) acupoints with sterilized electrode patches. The stimulation intensity and current intensity that gave the patient an effective pricking sensation ("Qi arrival") were maintained for 30 minutes. The stimulation method in the post-anesthesia care unit (PACU) was consistent with that before the operation.
  Arms: TEAS group
Device: Sham transcutaneous Electrical Acupoint Stimulation — Before the operation, disinfection patches with electrodes were applied to Zusanli (ST 36), Neiguan (PC 6), and Ciliao (BL 32) acupointst, but no electrical stimulation was conducted. The stimulation method in the post-anesthesia care unit (PACU) was the same as that before the operation.
  Arms: Sham group

SUMMARY:
The purpose of this clinical trial is to understand the effect of percutaneous acupoint electrical stimulation on postoperative gastrointestinal dysfunction. It will also investigate the safety of percutaneous acupoint electrical stimulation. The main questions that this trial aims to answer are:

Can percutaneous acupoint electrical stimulation alleviate postoperative gastrointestinal dysfunction? Through which mechanisms do they function?

Participants will:

Preoperatively, patients were either given or not given percutaneous acupoint electrical stimulation.

Record their symptoms and biological indicators within 5 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* BMI < 28 kg/m2
* ASA classification is I-III grade
* Preoperative pathological diagnosis is clear
* Laparoscopic surgury in urology under general anesthesia as a
* The patient has normal comprehension ability, and the patient or their family members can cooperate in filling out the questionnaire
* Voluntary to sign the informed consent form

Exclusion Criteria:

* Not meeting the above standards
* Having severe heart, lung or cerebrovascular diseases (such as severe coronary heart diseases, valve diseases, respiratory failure, cerebral hemorrhage, cerebral infarction, etc.)
* Having taken analgesic and gastrointestinal motility drugs before the operation
* Contraindications for TEAS (having electronic devices in the body， skin damage or infection at the stimulation site)
* Previous history of TEAS or electro-acupuncture treatment
* Previous history of long-term gastrointestinal motility disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
I-FEED(Intake, Feeling nauseated, Emesis, physical Exam, and Duration of symptoms)Score | Three days after the operation
  The I-FEED score consists of five aspects: eating, nausea, vomiting, physical examination, and duration of symptoms. The lowest score is 0 and the highest is 14. The higher the score, the worse the result. The normal I-FEED score is 0-2 points. Postoperative gastrointestinal intolerance (POGI) is 3-5 points, and Postoperative gastrointestinal dysfunction (POGD) is ≥ 6 points.

SECONDARY OUTCOMES:
The time of the first postoperative defecation and flatus expulsion | postoperative 3 days
The concentrations of motilin (MTL) | postoperative 5 days
Platelet/lymphocyte ratio (PLR) | postoperative 5 days
Visual analogue scale (VAS) Score | postoperative 5 days
  The VAS score refers to drawing a 10-cm scale on a piece of paper. One end of the scale is marked as 0, indicating no pain; the other end is marked as 10, indicating severe pain; the values in between represent different degrees of pain.
Quality-of-recovery 15 (Qor-15) Score | postoperative 1 day
  The QoR-15 includes 5 items related to physical comfort, 4 items regarding emotional state, 2 items concerning self-care ability, 2 items related to psychological support, and 2 items about pain. There are a total of 15 subjective parameters. Each item is scored on a scale of 0 to 10. The total score of QoR-15 ranges from 0 to 150. The higher the score, the better the condition.
miR-10b-5p | postoperative 5 days
Interleukin-6 (IL-6) | postoperative 5 days
Interleukin-10 (IL-10) | postoperative 5 days
Acetylcholine (Ach) | postoperative 5 days
Norepinephrine (NE) | postoperative 5 days

IPD SHARING:
Plan to Share IPD: No